CLINICAL TRIAL: NCT05464030
Title: A Phase I, Multicenter, Open-Label First in Human Study of Anti-CEACAM5 Antibody Drug Conjugate M9140 in Participants With Advanced Solid Tumors (PROCEADE-CRC-01)
Brief Title: Anti-CEACAM5 ADC M9140 in Advanced Solid Tumors (PROCEADE-CRC-01)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: EMD Serono Research & Development Institute, Inc. (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Organization: EMD Serono (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MS202329_0001; 2022-500508-23-00 (Other: EU CTIS)
Record Dates: First submitted 2022-07-15; First posted 2022-07-19 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab; Capecitabine; Fluorouracil; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part 1: M9140 (Experimental)
  Interventions: Drug: M9140
- Part 2A: M9140 (Experimental)
  Interventions: Drug: M9140
- Part 2B: M9140 (Experimental)
  Interventions: Drug: M9140
- Part 2C: M9140 + Bevacizumab +/-Capecitabine (Experimental)
  Interventions: Drug: M9140; Drug: Bevacizumab; Drug: Capecitabine
- Part 2D: M9140 + 5-fluorouracil + Folinic acid + Bevacizumab (Experimental)
  Interventions: Drug: M9140; Drug: 5-fluorouracil (5-FU); Drug: Folinic acid

INTERVENTIONS:
Drug: M9140 — M9140 will be administered at an escalated dose until Maximum tolerated dose (MTD) and/or a safe recommended Dose for Expansion (RDE) is determined in Part 1 of the study.
  Other Names: Precemtabart tocentecan
  Arms: Part 1: M9140
Drug: M9140 — M9140 will be further investigated in part 2 of the study and includes dose optimization, an alternative administration regimen and combination regimen.
  Other Names: Precemtabart tocentecan
  Arms: Part 2A: M9140; Part 2B: M9140; Part 2C: M9140 + Bevacizumab +/-Capecitabine; Part 2D: M9140 + 5-fluorouracil + Folinic acid + Bevacizumab
Drug: Bevacizumab — Bevacizumab will be administered intravenously as per standard of care.
  Arms: Part 2C: M9140 + Bevacizumab +/-Capecitabine
Drug: Capecitabine — Capecitabine will be administered orally as per standard of care.
  Arms: Part 2C: M9140 + Bevacizumab +/-Capecitabine
Drug: 5-fluorouracil (5-FU) — 5-FU will be administered intravenously as per standard of care.
  Arms: Part 2D: M9140 + 5-fluorouracil + Folinic acid + Bevacizumab
Drug: Folinic acid — Folinic acid will be administered intravenously as per standard of care.
  Arms: Part 2D: M9140 + 5-fluorouracil + Folinic acid + Bevacizumab

SUMMARY:
The purpose of this first-in-human study is to evaluate the safety, tolerability, pharmacokinetics, and preliminary clinical activity of M9140 in advanced solid tumors. This study contains 2 parts: Dose escalation (Part 1) and dose expansion (Part 2).

Study details include:

* Study Duration per participant: Approximately 4 months for Part 1 and 8 months for Part 2
* M9140 is not available through an expanded access program

ELIGIBILITY:
Inclusion Criteria:

* Participants with documented histopathological diagnosis of locally advanced or metastatic colorectal cancer (CRC), who were intolerant/refractory to or progressed after standard systemic therapies for the advanced/metastatic stage, if locally indicated and available to the participant. Participants with a known microsatellite instability high (MSI-H) status must have received treatment with an immune checkpoint inhibitor (if locally indicated and available) unless contraindicated.
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) below or equal to 1
* Participants with adequate hematologic, hepatic and renal function as defined in protocol
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* Participant has a history of malignancy within 3 years before the date of enrollment (exceptions are squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix, benign prostate neoplasm/hypertropia, or malignancy that in the opinion of the Investigator, with concurrence with the Sponsor's Medical Monitor, is considered cured with minimal risk of recurrence within 3 years)
* Participants with known brain metastases, except those meeting the following criteria: Brain metastases that have been treated locally and are clinically stable for at least 4 weeks prior to the start of treatment; No ongoing neurological symptoms that are related to the brain localization of the disease (sequelae that are a consequence of the treatment of the brain metastases are acceptable)
* Participants with diarrhea (liquid stool) or ileus Grade > 1
* Participants with active chronic inflammatory bowel disease (e.g., ulcerative colitis, Crohn's disease, intestinal perforation) and/or bowel obstruction
* Unstable angina, myocardial infarction, congestive heart failure (New York Heart Association [NYHA] >= II) or a coronary revascularization procedure within 180 days of study entry. Calculated QTc average (using the Fridericia correction calculation) of > 470 milliseconds (ms)
* Cerebrovascular accident/stroke (< 6 months prior to enrollment)
* Other protocol defined exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-08-04 (Actual); Primary Completion 2026-08-07 (Estimated); Study Completion 2026-08-07 (Estimated)

PRIMARY OUTCOMES:
Part 1: Number of Participants with Dose Limiting Toxicities (DLTs) and Adverse Events (AEs) | up to 4 months
Part 1: Recommended Dose Expansion (RDE) of M9140 | up to 4 months
Parts 2B, 2C and 2D: Number of Participants with Dose Limiting Toxicities (DLTs) and Adverse Events (AEs) | up to 8 months
Part 2A: Number of Participants with Adverse Events (AEs) | up to 8 months
Part 2A: Objective Response (OR) According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) as Assessed by Investigators | Time from first study treatment throughout the study duration until progressive disease or death up to approximately 8 months
Part 2A: Duration of Response (DoR) According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) as Assessed by Investigators | Time from first study treatment to planned assessment at approximately 8 months

SECONDARY OUTCOMES:
Parts 1, 2A, 2B, 2C and 2D: Pharmacokinetic (PK) Plasma Concentrations of M9140 | Part 1: Pre-dose up to 4 months; Part 2: Pre-dose up to 8 months
Parts 1, 2A, 2B, 2C and 2D: Number of Participants with Anti-Drug Antibodies (ADA) Against M9140 | Part 1: up to 4 months; Part 2: up to 8 months
Parts 1, 2A, 2B, 2C and 2D: Levels of Titers of Anti-Drug Antibody (ADA) Against M9140 | Part 1: up to 4 months; Part 2: up to 8 months
Parts 1 and 2A: Number of Participants with Clinically Significant Changes from Baseline in Triplicate 12-Lead Electrocardiogram (ECG) | Part 1: up to 4 months; Part 2: up to 8 months
Parts 1 and 2A: Change from Baseline in QTc (ΔQTc) Interval | Part 1: baseline, up to 4 months; Part 2: baseline up to 8 months
Parts 1, 2B, 2C: and 2D: Objective Response (OR) According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) as Assessed by Investigators | Time from first study treatment throughout the study duration until progressive disease or death up to approximately 4 months and 8 months
Parts 1, 2B, 2C and 2D: Duration of Response (DoR) According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) as Assessed by Investigator | Time from first study treatment to planned assessment at approximately 4 months and 8 months
Parts 2A, 2B, 2C and 2D: Time to Response | Time from first study treatment to planned assessment at approximately 8 months
Parts 1, 2A, 2B, 2C and 2D: Progression-free Survival (PFS) According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) as Assessed by Investigators | Time from first study treatment to planned assessment at approximately 4 months and 8 months
Part 2A: Overall Survival | Time from first study treatment to planned assessment at approximately 8 months
Part 2A: Number of Participants with Symptomatic Adverse Events (AEs) | up to 8 months
Parts 2A, 2B, 2C and 2D: Number of Participants with Disease Control | At Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — EMD Serono Research & Development Institute, Inc.
Locations (35):
- United States (6):
  - California Cancer Associates for Research & Excellence, Inc., Encinitas, California
  - California Cancer Associates for Research & Excellence, Inc., Fresno, California
  - Rhode Island Hospital, Providence, Rhode Island
  - Mary Crowley Cancer Research, Dallas, Texas
  - MD Anderson Cancer Center - Oncology, Houston, Texas
  - NEXT Oncology, San Antonio, Texas
- Canada (2):
  - The Ottawa Hospital Cancer Centre, Ottawa
  - University Health Network - Princess Margaret Cancer Centre, Toronto
- Japan (8):
  - National Cancer Center Hospital - Dept of Gastroenterology, Chūōku
  - National Cancer Center Hospital East, Kashiwa-shi
  - Saitama Cancer Center, Kitaadachi-gun
  - Cancer Institute Hospital of JFCR, Kōtoku
  - Aichi Cancer Center Hospital, Nagoya
  - Kindai University Hospital, Osakasayama-shi
  - Shizuoka Cancer Center, Sunto-gun
  - Kanagawa Cancer Center, Yokohama
- South Korea (7):
  - Kyungpook National University Chilgok Hospital, Daegu
  - National Cancer Center, Goyang-si
  - Seoul National University Bundang Hospital, Seongnam
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
- Spain (12):
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital HM Nou Delfos, Barcelona
  - Hospital Universitari Vall d'Hebron - VHIR, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - ICO l'Hospitalet - Hospital Duran i Reynals, L'Hospitalet de Llobregat
  - Centro Integral Oncologico Clara Campal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario Quironsalud Madrid - NEXT Oncology, Madrid
  - Complejo Hospitalario Universitario de Santiago, Santiago de Compostela
  - Hospital Universitario Virgen del Rocio, Seville

IPD SHARING:
Plan to Share IPD: No
We are committed to enhancing public health through responsible sharing of clinical trial data. Following approval of a new product or a new indication for an approved product in both the US and the European Union, the study sponsor and/or its affiliated companies will share study protocols, anonymized patient data and study level data, and redacted clinical study reports with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website https://bit.ly/IPD21

REFERENCES:
- [Result] Kopetz S, Boni V, Kato K, Raghav KPS, Vieito M, Pallis A, Habermehl C, Siddiqui A, Courlet P, Sloot W, Raab-Westphal S, Hart F, Rodriguez-Rivera I. Precemtabart tocentecan, an anti-CEACAM5 antibody-drug conjugate, in metastatic colorectal cancer: a phase 1 trial. Nat Med. 2025 Oct;31(10):3504-3513. doi: 10.1038/s41591-025-03843-z. Epub 2025 Jul 30. PMID 40739424
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS202329_0001
- See also: US Medical Information website, Medical Resources — https://medical.emdserono.com/en_US/home.html